CLINICAL TRIAL: NCT06098326
Title: Allogeneic Hematopoietic Cell Transplantation With Cyclophosphamide, Fludarabine, and Antithymocyte Globulin in Lower Risk Myelodysplastic Syndrome Phase 2 Extension Study
Brief Title: CyFluATG in Lower Risk MDS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Je-Hwan Lee, M.D. Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LRMDS_CyFluATG_2018
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Cyclophosphamide; fludarabine; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CyFluATG (Experimental): Patients who receive with cyclophosphamide, fludarabine, and antithymocyte globulin (CyFluATG) for allogeneic hematopoietic cell transplantation
  Interventions: Drug: cyclophosphamide, fludarabine, and antithymocyte globulin

INTERVENTIONS:
Drug: cyclophosphamide, fludarabine, and antithymocyte globulin — 1. Cyclophosphamide 50 mg/kg/day i.v. daily on days -3 and -2 (for 2 days)
  2. Fludarabine 30 mg/m2/day i.v. daily on days -7to -2 (for 6 days)
  3. Antithymocyte globulin (Thymoglobulin) 1.5 mg/kg/day (for HLA-matched sibling donor HCT) or 3.0 mg/kg/day (for other alternative donor HCT) i.v. daily on days -3 to -1 (for 3 days)

SUMMARY:
To evaluate the efficacy of the conditioning regimen with cyclophosphamide, fludarabine, and antithymocyte globulin (CyFluATG) for allogeneic hematopoietic cell transplantation (HCT) in patients with lower risk myelodysplastic syndrome (MDS). The efficacy of the treatment will be measured in terms of engraftment and non-relapse mortality (NRM).

DETAILED DESCRIPTION:
* This is a prospective, phase 2 extension study
* Conditioning regimen A. Cyclophosphamide 50 mg/kg/day i.v. daily on days -3 and -2 (for 2 days) B. Fludarabine 30 mg/m2/day i.v. daily on days -7to -2 (for 6 days) C. Antithymocyte globulin (Thymoglobulin) 1.5 mg/kg/day (for HLA-matched sibling donor HCT) or 3.0 mg/kg/day (for other alternative donor HCT) i.v. daily on days -3 to -1 (for 3 days) D. Methylprednisolone 2 mg/kg i.v. daily on days -4 to -1 (for 4 days)
* Harvest and infusion of donor hematopoietic cells A. Harvested peripheral blood mononuclear cells of donors via leukapheresis will be infused to recipients on day 0. Additional infusion on day 1 can be made based on the judgement of attending physician.
* GVHD prophylaxis A. Cyclosporine: 1.5 mg/kg i.v. every 12 hours beginning on day -1 and changed to oral dosing (with twice the i.v. dose) when oral intake is possible.

B. Methotrexate: 15 mg/m2 i.v. on day 1, and 10 mg/m2 i.v. on days 3 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lower risk MDS A. International prognosticscoring system (IPSS) ≤ 1.0 and B. Bone marrow blast percentage < 5% during the disease course before HCT
* Patients with appropriate hematopoietic cell donor A. HLA-matched sibling B. HLA-matched unrelated donor C. HLA-mismatched familial donor
* 18 years old or older, 70 years old or younger
* Adequate performance status (Karnofsky score of 70 or more)
* Adequate hepatic and renal function (AST, ALT, and bilirubin < 3.0 x upper normal limit, and creatinine < 2.0 mg/dL).
* Adequate cardiac function (left ventricular ejection fraction over 40% on heart scan or echocardiogram)
* Signed and dated informed consent must be obtained from both recipient and donor.

Exclusion Criteria:

* Presence of significant active infection
* Presence of uncontrolled bleeding
* Any coexisting major illness or organ failure
* Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible
* Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
engraftment and non-relapse mortality | 8 years
  To evaluate the efficacy of the conditioning regimen with cyclophosphamide, fludarabine, and antithymocyte globulin (CyFluATG) for allogeneic hematopoietic cell transplantation (HCT) in patients with lower risk myelodysplastic syndrome (MDS). The efficacy of the treatment will be measured in terms of engraftment and non-relapse mortality (NRM).

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea